CLINICAL TRIAL: NCT01133418
Title: Efficacy of a Cognitive Training Intervention for Children With ADHD
Brief Title: Cognitive Training Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Jeff Epstein, Principal Investigator, Children's Hospital Medical Center, Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: K24MH064478 (NIH)
Record Dates: First submitted 2010-05-17; First posted 2010-05-28 (Estimated); Results first posted 2017-05-01 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Training (Experimental): Computerized Progressive Attention Training
  Interventions: Other: Computerized Progressive Attention Training
- Non-progressive cognitive training (Sham Comparator): Children in the control condition will participate in the same tasks as children in the Intervention arm. They will experience the same number of blocks and trials of training as the intervention group. Further, their training will be conducted by the same set of trainers and for the same amount of time as the intervention group. However, children in the control group will remain at the lowest level for each CT task throughout training irrespective of performance.
  Interventions: Other: Sham Comparator Cognitive Training

INTERVENTIONS:
Other: Computerized Progressive Attention Training — Four comprehensive training tasks were developed and programmed based on expansions and modifications of various tasks that have been extensively investigated in the attention literature and are known to reflect primary attentional functions. Each task is discussed in detail in the Research Methods (section D.6.b). Briefly, they included a Continuous Performance Task, a Conjunctive Search Task, an Orienting and Flanker Task, and a Global-Local Task. All of the tasks were modified extensively from their original neuropsychological design to make them entertaining and stimulating enough for children to enjoy. Each task began at a relatively simple level of difficulty and gradually increased in difficulty across the training as children demonstrated proficiency according to reductions in RT variability
  Arms: Cognitive Training
Other: Sham Comparator Cognitive Training — Same tasks at Computerized Progressive Attention Training but the tasks do not progress in difficulty
  Arms: Non-progressive cognitive training

SUMMARY:
Currently, only two treatment modalities for pediatric attention deficit hyperactivity disorder (ADHD) are considered evidence-based: (1) pharmacological and (2) behavioral treatment. Recently, several studies have shown promising results suggesting efficacy for cognitive training interventions for children with ADHD. These interventions directly train cognitive function (i.e., attention, working memory) by having children practice cognitive skills using computerized tasks. In these studies, improvements related to the cognitive training intervention have been documented on neuropsychological tests, academic tasks, and parent ratings of children's ADHD behavior. Given the ubiquitous finding of increased reaction time (RT) variability among children with ADHD, the candidate worked with a group of developers to modify a cognitive training intervention to target RT variability. That is, train the children to be less variable in their responding. Initial clinical data from this intervention suggest that intervention exposure improves behavioral outcomes. However, an appropriate powered randomized clinical trial is necessary to experimentally demonstrate intervention efficacy.Sixty-four (64) children diagnosed with ADHD (either Predominantly Inattentive Type or Combined Type) will be randomly assigned to intervention or control conditions. Children in the intervention group will receive 8 weeks of the Computerized Progressive Attention Training (CPAT) intervention. Children in the control group will receive the CPAT intervention but there will be no progression in difficulty based on performance as in the intervention group. Children in both groups will be assessed pre-intervention and immediately after the 8-week training on neuropsychological, behavioral, and academic outcome measures. Hypothesis-driven data analyses will assess intervention efficacy.

Hypothesis #1: Children in the experimental group exposed to the CPAT intervention will show greater improvement from pre- to post-intervention on neuropsychological tests compared to children in the control group.

Hypothesis #2: Children in the experimental group exposed to the CPAT intervention will show greater improvement from pre- to post-intervention on parent and teacher behavioral ratings of ADHD behavior compared to children in the control group.

Hypothesis #3: Children in the experimental group exposed to the CPAT intervention will show greater improvement from pre- to post-intervention on academic outcomes compared to children in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Consent: The family must provide signature of informed consent by parents or legal guardians.
* Age at time of Screening: 7 to 12 years of age, inclusive.
* Gender: includes male and female children.
* ADHD Diagnostic Status: ADHD patients must meet DSM-IV criteria for ADHD-PIT or ADHD-CT subtype. Section D.4 below describes in detail the diagnostic process for arriving at diagnosis.
* Cognitive Functioning: IQ of greater than 80 as estimated by the Wechsler Abbreviated Scale of Intelligence.
* Learning Disability: Children must score above 75 on all three of the Wechsler Individual Achievement Test (WIAT) subtests (Reading, Spelling, Numerical Operations).
* School: Children must be enrolled in a school setting from which teacher ratings can be obtained.

Exclusion Criteria:

* Understanding Level. The patient and parent cannot understand or follow instructions given in the study.
* History of Psychiatric Medications: Children must not have taken psychiatric medications within the past month. In addition, the family must indicate that they do not plan on placing their child on medication for any psychiatric condition during the course of the study.
* Exclusionary Psychiatric Conditions: Children who meet diagnostic criteria on the K-SADS for OCD, any psychotic disorder, major depressive disorder or bipolar disorder will be excluded from participation.
* Developmental Disabilities. Patients will be excluded if they are deemed to be significantly developmentally delayed or have a pervasive developmental disorder. Developmental delay will be operationally defined as an IQ score below 80. A pervasive developmental delay will be defined as a T score above 65 on the Autism Composite Scale of the PDD Behavior Inventory.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2010-09; Primary Completion 2014-08 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Center for ADHD, Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cognitive Training | Non-progressive Cognitive Training
Started | 34 | 38
Completed | 29 | 32
Not Completed | 5 | 6
Not completed — Lost to Follow-up | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Training | Non-progressive Cognitive Training | Total
Number analyzed (Participants) | 34 | 38 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 34 | 38 | 72
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.71 (1.53) | 9.19 (1.84) | 8.98 (1.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 25 | 27 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 33 | 35 | 68
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 6 | 7 | 13
  White | 27 | 27 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 34 | 38 | 72

OUTCOME MEASURES:

1. Primary Outcome: Total ADHD Symptom Score From Vanderbilt ADHD Parent Rating Scale
Description: Total ADHD Symptom Score on the Parent Vanderbilt Rating Scales; range = 0-54; this score is computed by summing the 18 ADHD symptom items which are each rated on a 0-3 Likert scale (0="Never"; 1="Occasionally"; 2="Often"; 3="Very often"); higher scores indicate higher severity of ADHD symptoms.
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Training | Non-progressive Cognitive Training
Number analyzed (Participants) | 29 | 32
units on a scale | 27.00 (9.46) | 26.63 (10.08)
Statistical Analysis 1: Comparison: Cognitive Training vs Non-progressive Cognitive Training; Test type: Superiority or Other; p = .36, General Linear Model — a priori threshold for statistical significance was .05

2. Primary Outcome: Clinical Global Impression - Improvement
Description: Blinded ratings of clinical global impression - Improvement. Scale = 1 (Very Much Improved) - 7 (Very Much Worse) Lower scores represent more improvement.
Time Frame: 2 months
Population: One child in the Cognitive Training Group and one child in the Non-progressive Cognitive Training group were missing CGI data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Training | Non-progressive Cognitive Training
Number analyzed (Participants) | 28 | 31
units on a scale | 3.28 (.81) | 3.32 (.79)
Statistical Analysis 1: Comparison: Cognitive Training vs Non-progressive Cognitive Training; Test type: Superiority or Other; p = .86, General Linear Model

3. Secondary Outcome: Intra-individual Variability on Go/No-Go Task
Description: Standard deviation of reaction times for correct responses to Go trials on a Go/No-Go Task
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Cognitive Training | Non-progressive Cognitive Training
Number analyzed (Participants) | 27 | 27
milliseconds | 242.24 (100.55) | 236.60 (119.03)
Statistical Analysis 1: Comparison: Cognitive Training vs Non-progressive Cognitive Training; Test type: Superiority or Other; p = .79, General Linear Model

4. Secondary Outcome: Academic Improvement Measurement System - Web-based (AIMSWEB) Reading Score (Proportion Accurate)
Description: Number of words read correctly divided by number of words read (range = 0-1.0) Higher values represent better reading accuracy
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Training | Non-progressive Cognitive Training
Number analyzed (Participants) | 29 | 32
units on a scale | .97 (.03) | .97 (.04)
Statistical Analysis 1: Comparison: Cognitive Training vs Non-progressive Cognitive Training; Test type: Superiority or Other; p = .77, General Linear Model

ADVERSE EVENTS:
Arm/Group | Cognitive Training | Non-progressive Cognitive Training
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/38
Other Adverse Events (participants affected / at risk) | 0/34 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No